CLINICAL TRIAL: NCT03849898
Title: International, Multicenter, Prospective Registry to Collect Data in Patients 60 Years and Older Suffering From Mandibular Fractures
Brief Title: Patients 60 Years and Older Suffering From Mandibular Fractures Registry
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: MFx 60+_RP_v.1.0
Record Dates: First submitted 2019-02-15; First posted 2019-02-21 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Mandibular Fractures
Keywords: Fracture fixation; Surgical treatment; Non-Surgical treatment
MeSH Terms: conditions — Mandibular Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mandibular Fracture: Elderly patients of > 60 years who present a mandibular fracture
  Surgery or Non-surgical fracture treatment will be applied according to routine clinical practice
  Interventions: Procedure: Surgery; Other: Non-Surgical fracture treatment

INTERVENTIONS:
Procedure: Surgery — Surgical fracture treatment
  Other Names: Operative
Other: Non-Surgical fracture treatment — Non-Surgical fracture treatment

SUMMARY:
Approximately 200 of patients of 60 years or older who present a mandibular fracture will be enrolled in this registry. All patients will be treated and followed up according to the local standard (routine) of care at around 2 weeks, 6 weeks, 3 months and 6 months after treatment.

DETAILED DESCRIPTION:
Patients of 60 years or older who present a mandibular fracture will be enrolled in this registry. All patients will be treated (surgical or non-surgical) and followed up according to the local standard (routine) of care at around 2 weeks, 6 weeks, 3 months and 6 months after treatment.

Data collection will include patient and fracture details, treatment details, functional, clinical and patient-reported outcomes and anticipated or procedure- and implant-related adverse events (i.e. complications). Radiographs and/or other images (e.g. CT scan) taken as per standard of care will be collected within the registry.

Primary objectives are to obtain epidemiological data and describe the most common mandibular fracture patterns in older patients, to explore the relationship(s) between the treatment of mandibular fractures and its outcome in older patients, to identify risk factors and initiating factors of elderly related to mandible fracture events and to describe concomitant fractures associated with mandibular fractures in older patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years at the time of the injury
* Diagnosis of any kind of mandibular fracture
* Informed consent obtained, i.e.:

  * Ability to understand the content of the patient information/ informed consent form (ICF)
  * Willingness and ability to participate in the clinical investigation according to the Registry Plan (RP)
  * Signed and dated EC/IRB approved written informed consent OR For patients who are not able to provide independent written informed consent: Written consent provided according to defined and IRB/EC approved procedures

Exclusion Criteria:

* Patients with previous history of mandibular fractures or mandibular defects treated surgically
* Participation in any other medical device or medicinal product study within the previous months that could influence bone healing and the results of the present study in the opinion of the treating physician

Min Age: 60 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 60 years old with a mandibular fracture that requires treatment (either surgically or non-surgically)
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Patient-reported outcome | Baseline (preinjury)/ 2 weeks / 6 weeks / 3 months / 6 months
  Change in Geriatric/general Oral Self Assessment Index (GOHAI) over the follow up period:
  Self-reported measurement to describe three hypothetical dimensions 1) physical function, 2) psychosocial function and 3) pain and/or discomfort. It consisted of 12 items evaluated using a 5-point Likert from "never" to "always" in which higher scores indicated better outcomes.

OTHER OUTCOMES:
Occlusal Status | 2 weeks / 6 weeks / 3 months / 6 months
  Occlusion will be assessed without the use of dentures and classified follows:
  * Normal for the patient
  * Abnormal for the patient (multiple options possible)
    * Anterior open bite
    * Crossbite
    * Lateral open bite in the premolar area
    * Lateral open bite in the molar area
    * Deep bite: missing molar and/or pre-molar to support occlusion
    * Other
  * Not assessable (in case of edentulous patients or who use prosthesis)
Degree of malocclusion (if present) | 2 weeks / 6 weeks / 3 months / 6 months
  The thin-paper bite test will be used to evaluate the status of the occlusion. This test will be performed only if malocclusion is detected. Patients will be asked to close the mouth and bring teeth together while biting into a thin paper (<1mm). Deviations between opposite teeth greater than 1mm will be assessed as major, while deviations <1mm will be assessed as minor.
Mandibular dysfunction (Helkimo index) | 2 weeks / 6 weeks / 3 months / 6 months
  Evaluation by means Helkimo Index:
  1. Impaired range of movement (0 normal, 1 slight, 5 severely)
  2. Impaired temporomandibular joint function (0 smooth movement without joint sounds, 1 joint sounds in one or both joints, 5 locking and/or luxation of joint)
  3. Muscle pain (0 no tenderness, 1 tenderness to palpation in 1-3 palpation sites, 5 tenderness in 4 or more palpation sites)
  4. Temporomandibular joint pain (0 no tenderness, 1 tenderness to palpation laterally, 5 tenderness to palpation posteriority)
  5. Pain on movement (0 no pain, 1 pain one movement, 5 pain on two or more movements)
  Patients will be classified according to their score as follow:
  * 0 points, clinically symptom free
  * 1 - 4 points: mild dysfunction
  * 5 - 9 points: moderate dysfunction
  * 10 - 13 points: severe dysfunction
  * 15 - 17 points: severe dysfunction
  * 20 - 25 points: severe dysfunction
Mandibular Movements (mobility index) | 2 weeks / 6 weeks / 3 months / 6 months
  * Interincisal opening/maximal opening is defined as distance in millimeters between the edges of the incisors of the mandibular and the maxillary bone.
  * Lateral movements: With the mandible slightly open, it is defined as the distance in millimeters from the labioincisal embrasure between the central incisors to the labioincisal embrasure of the mandibular incisors
  * Protrusive movement: With the mandible slightly open, it is defined as the distance in millimeters between the incisal edges of the maxillary central incisor to the mandibular central incisor.
  Depending on the score, the mobility index will be calculated as follow:
  * 0 points: normal mandibular mobility
  * 1 - 4 points: slightly impaired mobility
  * 5 - 20 points: severely impaired mobility

CONTACTS AND LOCATIONS:
Overall Officials: Risto Kontio, Prof., Principal Investigator — Department of Oral and Maxillofacial Surgery, Helsinki University Hospital
Locations (24):
- United States (3):
  - UC Davis Health System, Sacramento, California
  - R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Harborview Medical Center, Seattle, Washington
- Helsinki University Hospital, Helsinki, Finland
- Germany (5):
  - University Hospital Freiburg, Freiburg im Breisgau
  - Medical Center Hamburg Eppendorf, Hamburg
  - Universitatsklinikum Marburg, Marburg
  - LMU - Klinikum der Universität München, München
  - Bundeswehrkrankenhauses Ulm, Ulm
- Hospital Sungai Buloh, Sungai Buloh, Malaysia
- Hospital General de Especialidades, Campeche, Mexico
- Erasmus MC, Rotterdam, Netherlands
- Spitalul Clinic Judeţean de Urgenţă "Sf. Apostol Andrei" Constanţa, Constanța, Romania
- Clinic for Maxillofacial Surgery, University of Belgrade, Belgrade, Serbia
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- King Edward VIII Hospital, Durban, South Africa
- Spain (3):
  - Hospital Vall d' Hebron, Barcelona
  - Hospital Puerta de Hierro, Madrid
  - Hospital Ramon y Cajal, Madrid
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- Universitaetsspital Basel, Basel, Switzerland
- National Cheng Kung University Hospital, Tainan, Taiwan
- Hospital Maciel de Montevideo, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Undecided